CLINICAL TRIAL: NCT00006345
Title: An Evaluation of Corticosteroid Pretreatment in Cutaneous T-Cell Lymphoma Patients Receiving Ontak (Denileukin Difitox)
Brief Title: Dexamethasone Followed by Denileukin Diftitox in Treating Patients With Persistent or Recurrent T-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ligand Pharmaceuticals (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Supportive Care
Other Study IDs: LIGAND-L4389-MR-9901; CDR0000068169 (Registry Identifier: PDQ (Physician Data Query)); NCI-V00-1614
Record Dates: First submitted 2000-10-04; First posted 2004-03-25 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2001-11

CONDITIONS: Drug/Agent Toxicity by Tissue/Organ; Lymphoma
Keywords: recurrent cutaneous T-cell non-Hodgkin lymphoma; drug/agent toxicity by tissue/organ; recurrent mycosis fungoides/Sezary syndrome
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Lymphoma; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome | interventions — denileukin diftitox; Dexamethasone

INTERVENTIONS:
Biological: denileukin diftitox
Drug: dexamethasone

SUMMARY:
RATIONALE: Denileukin diftitox may be able to deliver cancer-killing substances directly to T-cell lymphoma cells. Dexamethasone may decrease the side effects of denileukin diftitox.

PURPOSE: Phase II trial to study the effectiveness of dexamethasone in preventing side effects following treatment with denileukin diftitox in treating patients who have persistent or recurrent T-cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the potential benefit of dexamethasone administered prior to denileukin diftitox in terms of avoidance and/or reduction of hypersensitivity type reactions, flu-like symptom complex, and vascular leak syndrome side effects (adverse events) in patients with persistent or recurrent cutaneous T-cell lymphoma. II. Assess the response rate in terms of tumor burden reduction in these patients treated with this regimen. III. Determine the rate of patient withdrawal from the study due to adverse effects.

OUTLINE: This is an open label, multicenter study. Patients receive denileukin diftitox IV over 30-60 minutes on days 1-5. Patients also receive oral dexamethasone twice daily beginning 24 hours prior to and concomitantly with denileukin diftitox. Treatment continues every 3 weeks for at least 6 courses in the absence of disease progression or unacceptable toxicity. Patients are followed at 2 or 4 weeks.

PROJECTED ACCRUAL: Approximately 15-30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of persistent or recurrent cutaneous T-cell lymphoma (CTCL) and suitable for denileukin diftitox therapy

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Albumin at least 3.0 mg/dL Renal: Not specified Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception for at least 28 days prior to and during study No known hypersensitivity to denileukin diftitox or its components (e.g., diphtheria toxin, interleukin-2, or its excipients) or to dexamethasone No concurrent serious, uncontrolled infection that would preclude study

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics No prior denileukin diftitox (DAB389-interleukin-2) or DAB486-interleukin-2 No concurrent interferon Chemotherapy: No concurrent chemotherapy* No concurrent extracorporeal photochemotherapy* No concurrent systemic or combination cytotoxic chemotherapy No concurrent topical chemotherapy *For remission induction of CTCL Endocrine therapy: No other concurrent corticosteroids Radiotherapy: No concurrent electron beam radiotherapy and/or photophoresis Surgery: Not specified Other: At least 21 days since any prior anticancer therapy and recovered No other concurrent anticancer therapy for CTCL No concurrent experimental drugs or approved drugs tested in an investigational setting No concurrent topical therapy* No concurrent phototherapy* No concurrent cyclosporine No concurrent systemic retinoids *For remission induction of CTCL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-11; Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheila Stewart, MD, Study Chair — Ligand Pharmaceuticals
Locations (11):
- United States (11):
  - Veterans Affairs Medical Center - Miami, Miami, Florida
  - Rush Cancer Institute, Chicago, Illinois
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Arlington Cancer Center, Arlington, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas